CLINICAL TRIAL: NCT07167004
Title: Prompting a Switch From Refined Grains to Whole Grains in an Online Grocery Store Using Marketing Nudges and Financial Incentives
Brief Title: The GRoceries Aimed at Increasing Nutrition Study
Acronym: GRAINS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 858072; 2P30AG034546 (NIH)
Record Dates: First submitted 2025-07-25; First posted 2025-09-11 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes; Type II Diabetes Mellitus; Type II Diabetes; Pre-diabetes; Pre-diabetic; Pre-diabetic State; Type 2 Diabetes Mellitus (T2DM); Type 2 Diabetes Mellitus; Type 2 Diabetes (T2DM)
Keywords: chronic disease; diabetes; diabetes mellitus; type II diabetes; type 2 diabetes; pre-diabetes; prediabetes; whole grains; behavioral economics; marketing nudges; financial incentives; food is medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Chronic Disease; Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be informed that they will be randomly assigned to one of the three intervention arms, but they will not be told which group they are in. It will be necessary to omit these details so that participants will shop for their groceries as they would do in the real-world. The study team hopes this approach minimizes the chances that the participant will purchase foods that they think the study team wants them to purchase. Participants will be fully informed about the randomization process. To conceal the study's purpose, participants will be told that the study team is conducting consumer market research about online shopping experiences but will not be told the study team is specifically interested in understanding the effects of marketing and incentives on whole grain purchases. Participants will be fully debriefed at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Completion of weekly grocery shopping in a version of the study store without any interventions (i.e., without marketing nudges and financial incentives)
- Marketing Nudges Only (Experimental): Marketing nudges encouraging whole grain purchasing, including displaying whole grains (e.g., whole wheat bread, brown rice) at the top of the study's online grocery store, featuring whole grain banner displays, and offering product swaps to highlight whole grain alternatives
  Interventions: Behavioral: Marketing Nudges Only
- Marketing Nudges + Dynamically Adapted Financial Incentives (Experimental): Marketing nudges encouraging whole grain purchasing, including displaying whole grains (e.g., whole wheat bread, brown rice) at the top of the study's online grocery store, featuring whole grain banner displays, and offering product swaps to highlight whole grain alternatives, plus personalized financial incentives with individual incentive amounts optimized weekly based on prior whole grain purchasing behavior and engagement
  Interventions: Behavioral: Marketing Nudges + Dynamically Adapted Financial Incentives

INTERVENTIONS:
Behavioral: Marketing Nudges Only — Marketing nudges encouraging whole grain purchasing, including displaying whole grains (e.g., whole wheat bread, brown rice) at the top of the study's online grocery store, featuring whole grain banner displays, and offering product swaps to highlight whole grain alternatives
  Arms: Marketing Nudges Only
Behavioral: Marketing Nudges + Dynamically Adapted Financial Incentives — Marketing nudges encouraging whole grain purchasing, including displaying whole grains (e.g., whole wheat bread, brown rice) at the top of the study's online grocery store, featuring whole grain banner displays, and offering product swaps to highlight whole grain alternatives, plus personalized financial incentives with individual incentive amounts optimized weekly based on prior whole grain purchasing behavior and engagement
  Arms: Marketing Nudges + Dynamically Adapted Financial Incentives

SUMMARY:
Only 2% of Americans meet the recommended levels of whole grain consumption, despite its association with reduced risk of type 2 diabetes. This study aims to assess if consumers with prediabetes or type 2 diabetes can be encouraged to switch from buying refined grain products to whole grain products when shopping for groceries online. The study will use personalized marketing strategies, with or without discounts which adjust based on purchasing behavior, to promote whole grain consumption.

DETAILED DESCRIPTION:
The overall objective of this study is to determine if behaviorally informed marketing strategies or those same strategies plus dynamically adapted financial incentives can prompt consumers with prediabetes or diabetes to switch from refined to whole grain products when grocery shopping online. The specific aims of the study are:

Aim 1: To demonstrate the feasibility of conducting a randomized controlled trial (RCT) via an online grocery delivery platform and to refine mechanism-based marketing nudges and incentives based on user insights. The overall objective of this aim is to customize the online grocery store experience to align with the needs of the consumers while also supporting the objectives of the two intervention arms outlined in Aim 2. Customizations will include displaying whole grains (e.g., whole wheat bread, brown rice) at the top of the study's online grocery store, featuring whole grain banner displays, and offering product swaps to highlight whole grain alternatives. Additionally, the study team will ensure that all refined grain items have corresponding whole grain options, to the extent possible. To evaluate the platform's usability and gather insights for refining the interventions, the study team will recruit 9 participants to test the customized online grocery store. Participants will provide feedback on the online shopping environment and whole grain options in an end-of-study survey. This feedback will be used to refine the marketing nudge interventions for Aim 2.

Aim 2: To test whether behaviorally informed marketing strategies or those same strategies plus dynamically adapted financial incentives can prompt consumers with prediabetes or diabetes to switch from buying refined grain products to whole grain products when grocery shopping online. Enrolled participants will be randomized to one of three intervention arms: 1) control (no intervention), 2) marketing nudges, or 3) marketing nudges + dynamically adapted financial incentives. Participants will select groceries from the study's online grocery store, and the orders will be delivered to their homes via a third-party delivery service. The first two weeks will serve as a baseline period for data collection. Starting in Week 3, participants in intervention arms 2 and 3 will be exposed to marketing nudges promoting whole grains for 8 weeks. Participants in the third intervention arm will additionally receive personalized financial incentives with individual incentive amounts optimized weekly based on prior whole grain purchasing behavior and engagement. In a typical healthy eating incentive study, all participants would get the same incentive amount each week. An innovative aspect of this study is to dynamically adapt the incentive, so each person experiences a personalized offering of incentives each week based on their whole grain shopping habits in prior weeks. This means participants who did not buy a whole grain item in response to a smaller incentive in a prior week may receive a larger incentive than participants who did purchase whole grains when offered the smaller incentive. This will not be gameable since it will not be apparent to participants a priori. This approach enables us to mimic current retailer practices, rather than more outdated strategies that provide the same incentive weekly.

Aim 3: To examine whether whole grain purchasing behaviors have become habitual and persist after the marketing nudges and dynamically adapted financial incentives cease. The overall objective of this aim is to explore the potential for marketing strategies and dynamically adapted financial incentives to create lasting changes in grocery shopping habits, specifically by examining whether participants continue purchasing whole grain products once the intervention has ended. Participants will be followed for an additional 8 weeks post-intervention to track their online grocery shopping behavior in the absence of the marketing nudges and financial incentives. During this period, participants will continue to shop through the study's online grocery store and have their groceries delivered to them through a third-party delivery service. In addition, for the first 4 weeks of follow-up, they will continue to receive their weekly $10 incentive if they shop in the study's online grocery store. At the conclusion of the study, participants will receive a $25 incentive for completing a survey assessing the intervention's salience, their acceptance of whole grains, and any remaining barriers to switching to whole grains.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 - 70 years.
* Able to provide consent.
* Resident of Philadelphia, Bucks, Delaware, Chester, or Montgomery Counties in Pennsylvania.
* Consume <5 servings of whole grains per week.
* Use online grocery shopping at least once per month.
* Have access to a credit or debit card to pay for groceries purchased.
* Have reliable internet access.
* Speak English.
* Penn Medicine patient diagnosed with prediabetes or diabetes (identified using ICD-10 codes R73.03, E11).

Exclusion Criteria:

* Does not meet all the inclusion criteria.
* Not able to speak English.
* Not able to provide consent.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in calories purchased from products that are majority whole grains over time | 18 weeks
  The study team will use random-effects linear regression models to compare within-subject changes in the calories purchased from whole grains, adjusting for repeated measures, to examine trends over time.

SECONDARY OUTCOMES:
Change in calories purchased from products that are majority refined grains over time | 18 weeks
  The study team will use random-effects linear regression models to compare within-subject changes in the calories purchased from refined grains, adjusting for repeated measures, to examine trends over time.
Percent of cart spent on whole grains (total dollar on whole grains/cart total) | 18 weeks
  The study team will use mixed effects linear models with repeated observations to compare changes in this outcome.
Change in dollars spent on products that are majority whole grains over time | 18 weeks
  The study team will use mixed effects linear models with repeated observations to compare changes in this outcome.
Assessing whole and refined grain purchasing frequency | Assessed at baseline and in end-of-study survey (Week 18)
  The study team will assess the participant's self-reported purchasing frequency of different grain categories over the prior week, including rice and other cooked grains; oatmeal, grits, or other cooked cereal; cold cereal; bagels or English Muffins; breads or rolls; tortillas or wraps; pasta; and snacks (popcorn, crackers, granola bars). Response options include: never, 1 - 3 times per week, 4 - 6 times per week, 1 time per day, and 2 or more times per day.
Percentage of time grains were purchased as whole and refined grains | Assessed at baseline and in end-of-study survey (Week 18)
  The study team will assess how often each of the grain categories (i.e., rice and other cooked grains; oatmeal, grits, or other cooked cereal; cold cereal; bagels or English Muffins; breads or rolls; tortillas or wraps; pasta; and snacks [popcorn, crackers, granola bars]) were purchased as whole and refined grain products. Response options include: Almost never or never, About 25% of the time, About 50% of the time, About 75% of the time, and Almost always or always.
Assessing whole and refined grain consumption frequency | Assessed at baseline and in end-of-study survey (Week 18)
  The study team will assess the participant's self-reported consumption frequency of different grain categories over the prior week, including rice and other cooked grains; oatmeal, grits, or other cooked cereal; cold cereal; bagels or English Muffins; breads or rolls; tortillas or wraps; pasta; and snacks (popcorn, crackers, granola bars). Response options include: never, 1 - 3 times per week, 4 - 6 times per week, 1 time per day, and 2 or more times per day.
Percentage of time grains were consumed as whole and refined grains | Assessed at baseline and in end-of-study survey (Week 18)
  The study team will assess how often each of the grain categories (i.e., rice and other cooked grains; oatmeal, grits, or other cooked cereal; cold cereal; bagels or English Muffins; breads or rolls; tortillas or wraps; pasta; and snacks [popcorn, crackers, granola bars]) were consumed as whole and refined grain products over the prior week. Response options include: Almost never or never, About 25% of the time, About 50% of the time, About 75% of the time, and Almost always or always.
Amount of grains eaten at a time | Assessed at baseline and in end-of-study survey (Week 18)
  The study team will assess for each grain category how much was eaten at a time (i.e., in one sitting). Response options vary depending on the product.
Perception of whole grains: satisfaction with current whole grain consumption | Assessed at baseline and in end-of-study survey (Week 18)
  The outcome will be assessed with the following question: "I am satisfied with my current whole grain consumption" with response options structured as a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Perception of whole grains: beliefs about the impact of eating whole grains on health | Assessed at baseline and in end-of-study survey (Week 18)
  The outcome will be assessed with the following question: "I believe that eating whole grains positively impacts my health" with response options structured as a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Perception of whole grains: enjoyment of eating whole grains | Assessed at baseline and in end-of-study survey (Week 18)
  The outcome will be assessed with the following question: "I enjoy eating whole grains" with response options structured as a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Perception of whole grains: efforts to include whole grains in diet | Assessed at baseline and in end-of-study survey (Week 18)
  The outcome will be assessed with the following question: "I try to include whole grains in my diet" with response options structured as a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Perception of whole grains: confidence in ability to include whole grains in diet | Assessed at baseline and in end-of-study survey (Week 18)
  The outcome will be assessed with the following question: "I am confident I can include whole grains in my meals regularly" with response options structured as a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Perception of whole grains: capability of finding whole grains when shopping | Assessed at baseline and in end-of-study survey (Week 18)
  The outcome will be assessed with the following question: "I feel capable of finding whole grain options when grocery shopping" with response options structured as a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Perception of whole grains: whole grain affordability | Assessed at baseline and in end-of-study survey (Week 18)
  The outcome will be assessed with the following question: "Whole grain products are affordable for me" with response options structured as a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).
Perception of whole grains: whole grain taste | Assessed at baseline and in end-of-study survey (Week 18)
  The outcome will be assessed with the following question: "I find whole grain products to be tasty" with response options structured as a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Sophia V Hua, PhD, MPH, Principal Investigator — Department of Medical Ethics and Health Policy, Perelman School of Medicine
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be de-identified. De-identified IPD that underlie results in a publication can be requested by other researchers. The PI will review any and all requests to access the de-identified study data. SecureShare or PennBox, both secure methods to transfer files, will be used to transfer data.
Time Frame: One year after publication of the main trial results.
Access Criteria: The PI will review any and all requests to access the de-identified study data.